CLINICAL TRIAL: NCT06843746
Title: Comparison of Usability Satisfaction of the Newly Developed Low-cost Thermoplastic Splint and Commercial Thermoplastic Splint in Orthopedic Patients.
Brief Title: Comparison of Usability Satisfaction of the Newly Developed Low-cost Thermoplastic Splint and Commercial Thermoplastic Splint
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Komsak Sinsurin, Asst.Prof.Dr., Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MU-CIRB 2022/027.1002
Record Dates: First submitted 2025-02-19; First posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Usability Satisfaction
Keywords: Splinting Materials; Low temperature thermoplastic; Hand splint; Occupational Therapy

STUDY DESIGN:
Intervention Model Description: There are 2 groups: newly developed low-cost thermoplastic splint and commercial thermoplastic splint.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental)
  Interventions: Device: Newly developed low-cost thermoplastic
- Control group (Active Comparator)
  Interventions: Device: Commercial thermoplastic

INTERVENTIONS:
Device: Commercial thermoplastic — The participants received a commercial thermoplastic splint material for splint fabrication.
  Arms: Control group
Device: Newly developed low-cost thermoplastic — The participants received a newly developed low-cost thermoplastic splint material for splint fabrication.
  Arms: Experimental group

SUMMARY:
Low-temperature thermoplastic has been commonly used in the fabrication of hand splints. However, its high cost and limited accessibility pose challenges for both clinicians and clients. There is a need for innovative and cost-effective splinting materials that are convenient to use. This study aimed to investigate the satisfaction and opinions of patients regarding a newly developed low-cost thermoplastic material.

ELIGIBILITY:
Inclusion Criteria:

* Patient with musculoskeletal disorder
* Need to receive the splint from occupational therapist

Exclusion Criteria:

* History of neurological disorder
* Have the cognitive impairment
* Receive the splint already
* Have clinical diagnosis of the disease or symptoms that cannot use the splint

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 112 (Actual)
Dates: Start 2022-02-04 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction and opinions | After using the thermoplastic splint for 3 days
  An online questionnaire and Zoom Interview were utilized to collect the data on the satisfaction and opinions of orthopedic patients regarding the use of thermoplastic.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy, Mahidol University, Salaya, Changwat Nakhon Pathom, Thailand

IPD SHARING:
Plan to Share IPD: Undecided